CLINICAL TRIAL: NCT01584219
Title: The Role of Placental Myeloid Cells During Gestation, Labor and Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 0016-12HYMC
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-04

CONDITIONS: Congenital Anomaly of Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Women after cesarean section: Women after cesarean section
- pregnancy pathologies: pregnancy pathologies
- first/second trimester pregnancy
- Women after vaginal delivery: Women after vaginal delivery

SUMMARY:
Immature myeloid cells (IMCs) that are generated in the bone marrow, and differentiate into mature granulocytes, macrophages and dendritic cells (DCs) in the steady state. Recently, it was demonstrated that the IMC population expands in malignancy, both in animal models and in humans. These cells were described as immunosuppressants but have also been shown to promote tumor angiogenesis. Accordingly, IMCs were also found to take part in the burn injury wound healing process and other pathologies that involve angiogenesis. It was shown in the investigators' laboratory, that a very similar population of IMCs populates the mouse and human placenta, and that these cells actively promote angiogenesis.

Dendritic cells (DCs) that can differentiate from IMCs, are antigen presenting cells (APCs) that initiate and coordinate the innate and adaptive immune responses. DCs can take up a diverse array of antigens and present them to T cells as peptides bound to MHC products. These antigen-specific responses are critical for resistance to infection and tumors. Conversely, DCs have roles in autoimmunity, transplant rejection and immunological tolerance. In the reproductive system, DCs were shown to account for 5%-10% of all hematopoietic cells in the uterine decidua at the embryonic implantation site. They were shown to promote angiogenesis during early pregnancy, especially during implantation. Very little is known about their function in the placenta and in the latter part of pregnancy when significant angiogenesis takes part.

The investigators' preliminary mouse experiments and human data, demonstrate a shift in IMC/DC populations with the development of the placenta. The investigators hypothesize that this population shift may contribute to the labor and delivery process.

The investigators' aim is to understand the role of these myeloid cell populations during pregnancy, to characterize their phenotype and try to shed light on the cellular and molecular mechanisms of pregnancy complications, such as preeclampsia, pre-term labor, intrauterine growth restriction, etc.

DETAILED DESCRIPTION:
: Identification of proangiogenic myeloid cell populations in human placentas. Placental myeloid cells from different stages of pregnancy will be analyzed, using flow cytometry.

Aim 2: Characterization of the physiology of myeloid cells identified. Cells will be isolated, cultured and tested for proangiogenic properties using Matrigel plug assays, endothelial tube formation assays, etc. Immune tolerance will be analyzed in vitro using T cell proliferation studies, cytokine production, etc.

Aim 3: The role of placental myeloid cell populations in pathologies of pregnancy.

Placentas from human pregnancy pathologies that involve placental dysfunction, such as preeclampsia, pre-term labor, intrauterine growth restriction, will be analyzed using the methods mentioned above

ELIGIBILITY:
Inclusion Criteria:

* pregnant women

Exclusion Criteria:

* none

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Fainaru, PhD MD, Study Director — Technion, Israel Institute of Technology
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel